CLINICAL TRIAL: NCT06631937
Title: The Effect of Human Milk Oligosaccharides on Infant Gut Microbiota Modulation, Development of the Immune System and Health Later in Life: the BELIEF Study
Brief Title: HMOs on Infant Gut Microbiota Modulation and Development of the Immune System in Healthy Infants
Acronym: BELIEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other); Technical University of Denmark (Other); Chr Hansen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HND-IN-054
Record Dates: First submitted 2024-09-20; First posted 2024-10-08 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Healthy Infants
Keywords: infants; gastrointestinal microbiome; immune development; gastrointestinal well-being; infant formula fed

STUDY DESIGN:
Intervention Model Description: A randomized, placebo controlled trial of term infants with a 6 months intervention phase and 6 months short-term follow-up phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Human Milk Oligosaccharides (Experimental): Human Milk Oligosaccharides (HMO)
  Interventions: Other: Human Milk Oligosaccharides
- Placebo (Placebo Comparator): Identical commercial Infant Formula without human milk oligosaccharides, fed daily ad libitum from enrollement to 6 months of age
  Interventions: Other: Placebo
- Breastfed reference group (No Intervention)

INTERVENTIONS:
Other: Human Milk Oligosaccharides — Human Milk Oligosaccharides provided in a commercially available infant formula powder, fed daily ad libitum from enrollement to 6 months of age
  Arms: Human Milk Oligosaccharides
Other: Placebo — An identical commercially available infant formula powder without Human Milk Oligosaccharides, fed daily ad libitum from enrollement to 6 months of age
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn how a mixture of human milk oligosaccharides impacts the development of the infant microbiota, the immune maturation and how the interaction between the microbiota and immune maturation may impact both short and long term health of the infant.

The participants will:

* Consume the investigational products (active/placebo) for 6 months
* Legal guardians/parents to the participant to collect stool samples from the diapers at home
* Legal guardians/parents to the participant to report gastrointestinal symptoms, signs of infections in an electronic questionnaire
* Visit the clinic for checkups and dried blood sample collection

For reference, a group of breastfed infants will be included. They will undergo the same procedures apart from consuming the investigational product (active/placebo). 230 participants (115 in each intervention arm) will be randomized to an intervention and 104 participants will be recruited for the reference group, giving a total sample size of 334 participants.

The intervention trial will be reported in two steps, first step covering the intervention phase from birth to 6 months; and step two includes both the intervention phase (0-6 months) and the follow-up period from 6-12 months. Informed consents for the possibility to preform long-term follow-up will be obtained.

ELIGIBILITY:
Inclusion Criteria:

• All infants which parents has decided mode of feeding

Exclusion Criteria:

* Premature birth

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 334 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Total abundance of bifidobacteria at 3 months of age | Fecal samples collected at 3 months
  Abundance of fecal bifidobacteria measured by quantitative PCR

SECONDARY OUTCOMES:
Infant fecal pH at 3 months of age | Fecal samples collected at 3 months of age
  Fecal pH measured in fecal water at 3 months of age

OTHER OUTCOMES:
Infant growth | 1 week, 2 weeks, 1, 2, 3 and 6 months and 0-12 months
  Infant weight, length, and head circumference will be aggregated to determine infant growth status
Infant intestinal transit time | 9 months and 12 months
  Intestinal transit time estimated by sweet-corn transit time through the gastrointestinal tract
Frequency of Infections | 1 week, 2 weeks, 1, 2, 3 and 6 months
  Measured as episodes of respiratory and gastrointestinal infections within the first 6 months of age.
Infant crying and fussing | 1 week, 2 weeks, 1, 2, 3 and 6 months
  Measured as frequency/duration of crying and fussing assessed as parent-reported in the Infant Health Questionnaire
General health status of infants | 0-12 months
  General health status measured as number of health care visits and illness diagnosis
Infant stool frequency | 1 week, 2 weeks, 1, 2, 3 and 6 months
  Changes in stool frequency and consistency measured from birth through to 6 months of age assessed as parent-reported in the Infant Health Questionnaire
Infant fecal immunoglobulins | 1 week, 2 weeks, 1, 2, 3 and 6 months and 0-12 months
  Changes in fecal immunoglobulins from infant fecal samples
Infant blood immunoglobulins | 3, 6 and 12 months
  Changes in immunoglobulins measured in dried blood spots
Characterization of Infant gut metabolome | 1 week, 2 weeks, 1, 2, 3, 6, 9 and 12 months
  Characterization and changes in the Infant fecal metabolome as assessed by targeted and untargeted metabolomics
Characterization of the Infant blood metabolome | 3, 6 and 12 months
  Characterization and changes of the Infant blood metabolome as assessed by targeted and untargeted metabolomics from dried blood spots
Characterization of the Infant gut microbiome composition | 1 week, 2 weeks, 1, 2, 3, 6, 9 and 12 months
  Changes in gut microbiome composition analyzed by DNA/RNA sequencing of fecal samples.
Characterization of Infant blood cytokine profiles | 3, 6 and 12 months
  Changes in pro-inflammatory and anti-inflammatory cytokines profiles from dried blood spots
Characterization of Infant fecal cytokines profiles | 1 week, 2 weeks, 1, 2, 3 and 6 months and 0-12 months
  Changes in pro-inflammatory and anti-inflammatory cytokines profiles measured in fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Lars H Pedersen, Professor, PhD, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No